CLINICAL TRIAL: NCT05009160
Title: DreaMS - Development of Digital Biomarkers in Multiple Sclerosis - Validation Study 1
Brief Title: DreaMS - Validation Study 1
Status: Recruiting | Type: Observational
Sponsor: Research Center for Clinical Neuroimmunology and Neuroscience Basel (Other)
Collaborators: University Hospital, Basel, Switzerland (Other); University of Basel (Other); Innosuisse - Swiss Innovation Agency (Other); Novartis Pharmaceuticals (Industry); Hoffmann-La Roche (Industry); Indivi AG (Industry)
Responsible Party: Sponsor
Other Study IDs: DreaMS_2021VS1; SNCTP000004678 (Registry Identifier: Swiss National Clinical Trials Portal)
Record Dates: First submitted 2021-07-23; First posted 2021-08-17 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-11

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Digital Biomarker
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with Multiple Sclerosis (PwMS): PwMS will download the Indivi platform App which contains the dreaMS App and will follow the study schedule.
  Interventions: Device: dreaMS App R2.1
- Healthy Control Persons (HC): HC will download the Indivi platform App which contains the dreaMS App and will follow the same study schedule as PwMS.
  Interventions: Device: dreaMS App R2.1

INTERVENTIONS:
Device: dreaMS App R2.1 — The Healios+Me platform App which contains the dreaMS App will be downloaded by all participants and all participants (PwMS and HC) will follow the same schedule

SUMMARY:
Multiple Sclerosis (MS) is a chronic inflammatory disease of the central nervous system (CNS) causing focal lesions of demyelination and diffuse neurodegeneration in the grey and white matter of the brain and spinal cord, leading to physical and cognitive disability. The scientific community and patients are in need for new and more reliable biomarkers, especially biomarkers of disease progression in order to adapt therapeutic approaches on an individual level. Digital biomarkers have the potential to fill this gap allowing for quasi-continuous measures that might be more informative than episodically collected conventional data concerning the impact of the disease on activities of daily living.

Using app-based challenges, continuous monitoring and surveys the Investigators aim to obtain data that can be used as digital biomarkers (DB). These digital biomarkers will provide more granular and precise assessments, thus complementing traditional diagnostic measures and techniques. After a first feasibility study (ClinicalTrials.gov: NCT04413032) a number of digital biomarkers have been identified as reliable, reproducible and meaningful to PwMS and are therefore being validated in a bigger cohort of PwMS with a longer follow-up within this validation study 1. Those digital biomarkers will be compared to state-of-the-Art clinical, imaging and body fluid assessment.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a chronic inflammatory disease of the central nervous system (CNS) causing focal lesions of demyelination and diffuse neurodegeneration in the grey and white matter of the brain and spinal cord, leading to physical and cognitive disability. Currently there is a limited number of relevant biomarkers available in persons with MS (PwMS), such as clinical, imaging or biological measures. Patient history and neurologic examination in combination with magnetic resonance imaging (MRI), evoked potentials and analysis of serum and cerebrospinal fluid (CSF) are the gold standard of diagnosis and mainly patient history, neurologic examination and MRI are used for patient monitoring. However, their prognostic value on a patient level is still very limited. Therefore, the scientific community and patients are in need for new and more reliable biomarkers, especially biomarkers of disease progression in order to adapt therapeutic approaches on an individual level. Digital biomarkers have the potential to fill this gap allowing for quasi-continuous measures that might be more informative than episodically collected conventional data concerning the impact of the disease on activities of daily living.

The Investigators have developed the Healios+Me platform App which contains the dreaMS App and serves as a data collection, communication and management platform using data collected through the patients' mobile devices (smartphone and wearables). Using the dreaMS app-based challenges, continuous monitoring and surveys the Investigators aim to obtain data that can be used as digital biomarkers (DB). These digital biomarkers will provide more granular and precise assessments, thus complementing traditional diagnostic measures and techniques. After a first feasibility study (ClinicalTrials.gov: NCT04413032) a number of digital biomarkers have been identified as reliable, reproducible and meaningful to PwMS and are therefore being validated in a bigger cohort of PwMS with a longer follow-up within this validation study 1. Those digital biomarkers will be compared to state-of-the-Art clinical, imaging and body fluid assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Diagnosed with MS according to the revised McDonald criteria 2017, all clinical forms inclusive (CIS, RRMS, SPMS, PPMS), for PwMS only
* In possession of a Healios+Me App compatible smartphone (iOS/Android)
* Corrected close visual acuity of ≥0.5
* Hand motor skills sufficient for using a smartphone
* Ability to follow the study procedures
* Informed Consent as documented by signature

Exclusion Criteria:

* Being diagnosed with MS or other disease affecting neurological and cognitive functions, for HC only
* Other clinically significant concomitant disease states (e.g., renal failure, severe hepatic dysfunction, severe/unstable cardiovascular disease, progressive cancer, etc.)
* Known or suspected non-compliance, drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants of this study will be recruited from the outpatient department of the MS Center Basel at the University Hospital Basel.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Correlation of the digital features with the respective measurements of the clinical reference tests | Baseline to last visit (year two)
  Spearman correlation coefficients higher than 0.4 (lower bound of 95% confidence interval) are considered relevant. All scheduled pairs of measurements collected during the study will be used. As the yearly observations of a patient are not independent, standard conﬁdence intervals cannot be used. Therefore, a bootstrap approach will be used to determine a 95% conﬁdence interval for the Spearman correlations (where data will be resampled on the patient level).
The ability of measurements of the changes in the digital biomarkers over the two-year follow-up to predict worsening in the clinical reference test over the same period expressed as binary variables | Measurements at baseline and after two years
  The change of the digital biomarker over two years allows to distinguish patients experiencing a relevant worsening in the corresponding reference test over the same period from those who do not with an area under the receiver operating characteristic curve (AUC) larger than 0.6 (lower bound of 95% confidence interval).

CONTACTS AND LOCATIONS:
Overall Officials: Ludwig Kappos, Study Director — Research Center for Clinical Neuroimmunology and Neuroscience Basel; Jannis Müller, Principal Investigator — RC2NB and Department of Neurology, University Hospital of Basel, Switzerland
Locations (6):
- Switzerland (6):
  - Neurozentrum, Kantonsspital Aarau, Aarau, Switzerland
  - Department of Neurology, CHUV Lausanne, Lausanne, Switzerland
  - Centro Sclerosi Multipla, Ospedale Regionale di Lugano, Lugano, Switzerland
  - Klinik für Neurologie, Kantonsspital St. Gallen, Sankt Gallen, Switzerland
  - Klinik für Neurologie, Universitätsspital Zürich, Zurich, Switzerland
  - MS Center, Department of Neurology University Hospital Basel, Basel

IPD SHARING:
Plan to Share IPD: Undecided